CLINICAL TRIAL: NCT00730028
Title: Randomized, Double-Blind Trial of Clindamycin, Trimethoprim-Sulfamethoxazole, or Placebo for Uncomplicated Skin and Soft Tissue Infections Caused by Community-Associated Methicillin-Resistant Staphylococcus Aureus
Brief Title: Uncomplicated Skin and Soft Tissue Infections Caused by Community-Associated Methicillin-Resistant Staphylococcus Aureus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-0051; UCSF CA-MRSA
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2015-04

CONDITIONS: Staphylococcal Infection
Keywords: Methicillin-resistant Staphylococcus aureus (MRSA), cellulitis, abscess, children, elderly
MeSH Terms: conditions — Staphylococcal Infections; Cellulitis; Abscess | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Limited Abscess (Experimental): Limited abscess with or without cellulitis less than or equal to 5 cm in diameter will be randomized to receive a 10-day course a) TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children; or b) CLINDA 300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children; or c) placebo two capsules three times daily.
  Interventions: Drug: Trimethoprim-sulfamethoxazole; Other: Placebo; Drug: Clindamycin
- Cellulitis or Larger Abscess (Experimental): Subjects with cellulitis only or abscess > 5 cm in diameter, or with 2 or more sites of skin infection will be randomized to receive a 10-day course a) TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children; or b) CLINDA300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children.
  Interventions: Drug: Trimethoprim-sulfamethoxazole; Drug: Clindamycin

INTERVENTIONS:
Drug: Trimethoprim-sulfamethoxazole — Trimethoprim-sulfamethoxazole (TMP-SMX) will be administered orally at a dose of 160 mg TMP and 800 mg SMX (as 2 single strength over encapsulated tablets) twice daily (adult or child > 40 kg dose) or 8-10 mg TMP, 40-50 mg SMX per kg daily, divided into 2 daily doses (child < 40 kg dose). Study drug will be administered for 10 days.
Other: Placebo — Placebo capsules will be identical in appearance to the CLINDA and TMP-SMX. Administered 3 times daily for 10 days.
  Arms: Limited Abscess
Drug: Clindamycin — CLINDA (adult dose of 300 mg three times daily; pediatric dose of 25-30 mg/kg/day divided three times daily up to a maximum dose of 900 mg/day). Study drug will be administered for 10 days.

SUMMARY:
The purpose of this clinical trial is to evaluate 2 different antibiotics, drugs that fight bacteria, [clindamycin (CLINDA) and trimethoprim-sulfamethoxazole (TMP-SMX)] and wound care for the outpatient management of uncomplicated skin and soft tissue infections (uSSTIs) in children and adults. The study will occur in areas where community associated methicillin-resistant Staphylococcus (S.) aureus are common. S. aureus is a type of bacteria. A total of 1310 volunteers, greater than or equal to 6 months of age and adults 85 years or younger, non-immunocompromised, with uSSTIs (in particular abscess and/or cellulitis) will be enrolled in this study. Subjects will be treated with one of the following: CLINDA, TMP-SMX, or placebo (contains no medication). Volunteers will be grouped based on the presence of cellulitis or abscess, whether the abscess can be surgically drained, and its size. The subject participation duration for this study is about 6 weeks.

DETAILED DESCRIPTION:
Clinical practice in the treatment of community-onset skin and soft tissue infections (SSTI) has not kept pace with the emergence of methicillin-resistant Staphylococcus aureus (MRSA) in the community. This clinical trial will evaluate clindamycin (CLINDA) and trimethoprim-sulfamethoxazole (TMP-SMX) and wound care for the outpatient management of uncomplicated skin and soft tissue infection (uSSTI) in 3 metropolitan areas, Chicago, Los Angeles, and San Francisco, cities with high prevalence of community acquired (CA)-MRSA. This is a phase IIb multicenter, stratified, randomized, double-blind trial in which enrolled subjects with abscess or cellulitis will be treated with CLINDA, TMP-SMX, or placebo. Participants will include 1310 non-immunocompromised out-patients age 6 months to 85 years with SSTIs not requiring hospital admission. Subjects will undergo a screening/baseline evaluation, including determination of presence and size of abscess and/or presence of cellulitis. Subjects will then be randomized to receive treatment with either CLINDA, TMP-SMX, or placebo depending on whether they have: a larger drainable abscess, defined as greater than 5 cm in diameter in adults and as greater than 3 cm in diameter for ages 6-11 months, greater than 4 cm for ages 1-8 years, and greater than 5 cm for age 9 years and older; a limited drainable abscess, defined as less than or equal to 5 cm for adults and as less than or equal to 3 cm for ages 6-11 months, less than or equal to 4 cm for ages 1-8 years, and less than or equal to 5 cm for age 9 years and older; or cellulitis or erysipelas only. If the diameter of the abscess greater than 5 cm (smaller for children depending on age) or 2 or more sites of skin infection are present the subject will be randomized (1:1) to 10 days of therapy with TMP-SMX or CLINDA. If the diameter of the abscess less than or equal to 5 cm (smaller for children depending on age) then the subject will be randomized (1:1:1) to TMP-SMX, CLINDA or placebo for 10 days. Subjects with cellulitis or erysipelas only will be randomized (1:1) to TMP-SMX or CLINDA for 10 days. Subjects will be provided study drug, instructed in its use, and scheduled for 4 follow-up visits including: wound check (24-48 hours after enrollment); end of therapy (48 hours after completion of therapy); test of cure (7-10 days after completion of therapy); and a final visit at one month after completion of therapy. The primary objectives of this study are: to compare the cure rate of CLINDA to that of TMP-SMX for the treatment of patients with cellulitis or larger abscess at the Test of Cure (TOC) visit and to compare the cure rate of CLINDA, TMP-SMX, and placebo, each in conjunction with surgical drainage for the treatment of subjects with limited abscess at the TOC visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 85 years.
* Able to complete the informed consent process or, if a minor, a parent or guardian who is able to complete the informed consent process; an assent form also will be completed for children age 7 and older.
* Willing and able to complete the study protocol, study-related activities, and visits.
* Diagnosis of uncomplicated skin and soft tissue infection (uSSTI), either cellulitis (defined as an inflammation of skin and associated skin structures) or abscess (defined as a circumscribed collection of pus), evidenced by at least 2 of the following localized signs or symptoms on the skin for at least 24 hours:

  1. Erythema
  2. Swelling or induration
  3. Local warmth
  4. Purulent drainage
  5. Tenderness to palpation or pain
* Able to take oral antibiotic therapy, either in pill or suspension form.

Exclusion Criteria:

* Hospital in-patient.
* Hospitalization within the prior 14 days.
* Residence in a long-term skilled nursing facility.
* Requirement for hospitalization for skin infection or other condition.
* Previous enrollment in this protocol.
* Participation in another clinical trial within the previous 30 days.
* Superficial skin infection only, including:

  1. Impetigo
  2. Ecthyma
  3. Folliculitis
  4. Infections that have a high cure rate after surgical incision alone (such as isolated furunculosis) or after topical or local measures
* Unstable psychiatric or psychological condition rendering the subject unlikely to be cooperative or to complete study requirements.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with the adherence or subject compliance with study requirements.
* Systolic blood pressure > 180 mm Hg.
* Systolic blood pressure (SBP) less than an age-specific critical value:

  1. Age 6 - 11 months: < 70 mm Hg
  2. Age 1 to 8 years: < 80 mm Hg
  3. Age 9 to 17 years: < 90 mm Hg
  4. Age greater than or equal to 18 years: < 90 mm Hg
* Heart rate less than 45 beats per minute (BPM).
* Heart rate greater than an age-specific critical value:

  1. Age 6 - 11 months: > 140 BPM
  2. Age 1 to 8 years: > 120 BPM
  3. Age 9 to 17 years: > 120 BPM
  4. Age greater than or equal to 18 years: > 120 BPM.
* Oral temperature (or equivalent rectal, tympanic membrane, axillary) less than 35.5 degrees Celsius (95.9 degrees Fahrenheit).
* Oral temperature (or equivalent rectal, tympanic membrane, axillary) greater than age-specific critical value:

  1. Age 6 - 11 months: > 38.0 degrees Celsius (100.4 degrees Fahrenheit)
  2. Age 1 to 8 years: > 38.5 degrees Celsius (101.3 degrees Fahrenheit)
  3. Age 9 to 17 years: > 38.5 degrees Celsius (101.3 degrees Fahrenheit)
  4. Age greater than or equal to 18 years: > 38.5 degrees Celsius (101.3 degrees Fahrenheit).
* Documented human or witnessed animal bite in the past 30 days at the site of infection.
* Systemic antibacterial therapy with antistaphylococcal activity within the prior 14 days.
* The following concomitant medications: warfarin, phenytoin, methotrexate, rosiglitazone or sulfonylureas and systemically administered antibacterial agents with activity against staphylococci.
* Diagnosed or suspected disseminated or severe Staphylococcus aureus or group A streptococcal (GAS) infection, including lymphangitic spread of skin infection, septicemia, bacteremia, pneumonia, endocarditis, osteomyelitis, septic arthritis, gangrene, necrotizing fasciitis, myositis, or other serious infections.
* Infection at an anatomical skin site requiring specialized management or specialized antimicrobial therapy, including:

  1. Periauricular or orbital infection
  2. Perirectal infection
  3. Suspected deep space infection of the hand or foot
  4. Genital infection
  5. Mastitis
  6. Bursitis
* Radiographic evidence or suspicion of gas in the tissue or foreign body infection (note: radiography is not required for screening and can be performed at the discretion of the treating physician).
* Gastrointestinal symptoms such as nausea, vomiting, or diarrhea of a severity that would preclude consumption of oral antibiotics.
* Hypersensitivity or history of allergic reaction to study drug.
* History of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Third trimester pregnancy: pregnant women must have gestational age estimated by an objective means, e.g. ultrasound, fundal height, and women who are within 4 weeks of the third trimester of pregnancy, defined as week 27 of pregnancy, are not eligible.
* Currently breast feeding.
* Severe or morbid obesity with a body mass index (BMI) >40 kg/m^2.
* Complicated skin or soft tissue infection, such as:

  1. Catheter or catheter site infection within 30 days of placement
  2. Surgical site infection
  3. Known or suspected prosthetic device infection
  4. Suspected Gram-negative or anaerobic pathogen
  5. Unusual exposure history (e.g., underwater injury, fish-tank exposure, heavy soil exposure, etc)
  6. Infection at the site of an area of underlying skin disease such as chronic eczema, psoriasis, atopic dermatitis, or chronic venous stasis
* History of underlying immunocompromising condition or immunodeficiency, for example:

  1. Diabetes mellitus
  2. Chronic renal failure, creatinine clearance <30 ml/min
  3. Renal dialysis within the past 180 days
  4. Human immunodeficiency virus (HIV)-positive with either cluster of differentiation (CD)4 count <200 or <4 percent CD4 in the past 180 days or HIV-positive and no documented CD4 count in the past 4 months
  5. Organ or bone marrow transplantation (ever), immunosuppressive therapy within the past 180 days, severe liver disease
  6. Other serious underlying disease, as determined by the treating physician or the investigator

Ages: 6 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1310 (Actual)
Dates: Start 2009-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - San Francisco General Hospital - Infectious Diseases, San Francisco, California
  - Harbor UCLA Medical Center - Medicine - Infectious Diseases, Torrance, California
  - Morehouse School of Medicine - Morehouse Medical Associates - Atlanta, Atlanta, Georgia
  - The University of Chicago - Comer Children's Hospital - Infectious Diseases, Chicago, Illinois
  - Washington University School of Medicine in St. Louis - Infectious Diseases, St Louis, Missouri
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee

REFERENCES:
- [Result] Miller LG, Daum RS, Creech CB, Young D, Downing MD, Eells SJ, Pettibone S, Hoagland RJ, Chambers HF; DMID 07-0051 Team. Clindamycin versus trimethoprim-sulfamethoxazole for uncomplicated skin infections. N Engl J Med. 2015 Mar 19;372(12):1093-103. doi: 10.1056/NEJMoa1403789. PMID 25785967
- [Derived] Daum RS, Miller LG, Immergluck L, Fritz S, Creech CB, Young D, Kumar N, Downing M, Pettibone S, Hoagland R, Eells SJ, Boyle MG, Parker TC, Chambers HF; DMID 07-0051 Team. A Placebo-Controlled Trial of Antibiotics for Smaller Skin Abscesses. N Engl J Med. 2017 Jun 29;376(26):2545-2555. doi: 10.1056/NEJMoa1607033. PMID 28657870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were non-immunocompromised out-patients age 6 months to 85 years with SSTIs not requiring hospital admission were recruited across 6 sites from communities with an anticipated prevalence of community-associated MRSA. Participants were enrolled between April 13, 2009 and January 13, 2015
Groups:
- Cellulitis or Larger Abscess - Clindamycin: Participants with cellulitis only or abscess > 5 cm in diameter in adults and children age 9 years and older, > 4 cm in diameter in children age 1 to 8 years, or > 3 cm in diameter in children age 6 to 12 months, or with 2 or more sites of skin infection were treated with CLINDA300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children.
- Cellulitis or Larger Abscess - TMP-SMX: Participants with cellulitis only or abscess > 5 cm in diameter in adults and children age 9 years and older, > 4 cm in diameter in children age 1 to 8 years, or > 3 cm in diameter in children age 6 to 12 months, or with 2 or more sites of skin infection were treated with TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children.
- Limited Abscess - Clindamycin: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter in adults and children age 9 years and older, < 4 cm in diameter in children age 1 to 8 years, or < 3 cm in diameter in children age 6 to 12 months were treated with CLINDA300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children.
- Limited Abscess - TMP-SMX: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter in adults and children age 9 years and older, < 4 cm in diameter in children age 1 to 8 years, or < 3 cm in diameter in children age 6 to 12 months were treated with TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children.
- Limited Abscess - Placebo: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter in adults and children age 9 years and older, < 4 cm in diameter in children age 1 to 8 years, or < 3 cm in diameter in children age 6 to 12 months were treated with placebo three times daily.
Period: Overall Study
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Started | 264 | 260 | 266 | 263 | 257
Completed | 204 | 194 | 221 | 207 | 175
Not Completed | 60 | 66 | 45 | 56 | 82
Not completed — Adverse Event | 23 | 26 | 16 | 20 | 43
Not completed — Lost to Follow-up | 13 | 26 | 22 | 26 | 25
Not completed — Protocol Violation | 6 | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 4 | 5 | 9
Not completed — Physician Decision | 3 | 3 | 2 | 3 | 2
Not completed — Treatment Failure | 5 | 5 | 0 | 0 | 1
Not completed — Randomization Error | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the protocol are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo | Total
Number analyzed (Participants) | 264 | 260 | 266 | 263 | 257 | 1310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 81 | 74 | 101 | 91 | 89 | 436
  Between 18 and 65 years | 181 | 184 | 164 | 169 | 166 | 864
  >=65 years | 2 | 2 | 1 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (17.2) | 27.5 (16.9) | 24.8 (17.8) | 25.6 (18.1) | 26.2 (18.7) | 27.1 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 121 | 126 | 111 | 101 | 588
  Male | 135 | 139 | 140 | 152 | 156 | 722
Region of Enrollment [Number; unit: participants]
  United States | 264 | 260 | 266 | 263 | 257 | 1310

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Cure, Defined as Absence of Clinical Failure, in the Evaluable Population.
Description: Clinical failure is defined as the occurence of any of the following:
  1. Lack of resolution at the Test of Cure (TOC) visit in any or all of the following: erythema, tenderness, purulent drainage, swelling, and local warmth. Erythema or tenderness that was considered due the surgical therapy itself (incision and drainage), was not considered to be indicative of clinical failure.
  2. Occurrence of a SSTI at another site other than the site(s) under study.
  3. Intolerance of study medication or a treatment-limiting adverse reaction necessitating discontinuation of study drug within the first 48 hours.
  4. Administration of other antimicrobial therapy for treatment of a SSTI at any time through the TOC visit.
  5. Unplanned surgical procedure for the infection under study at any time through the TOC visit.
  6. Hospitalization for treatment of active or invasive infection at any time through the TOC visit.
Time Frame: Test of cure (TOC) (7-10 days after completion of therapy)
Population: The efficacy evaluable population was comprised of all participants who had outcomes determined at the Test of Cure (TOC) visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 237 | 229 | 238 | 232 | 220
percentage of participants | 89.5 [85.2 to 93.7] | 88.2 [83.7 to 92.7] | 92.9 [89.3 to 96.4] | 92.7 [89.0 to 96.3] | 80.5 [74.8 to 86.1]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; Primary null hypothesis: Clindamycin and TMP-SMX have equal rates of cure in the treatment of cellulitis/larger abscess at the Test of Cure (TOC) visit; Test type: Superiority or Other; p = 0.7688, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-7.6 to 5.1] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; Primary null hypothesis: After successful surgical drainage, placebo, Clindamycin, and TMP-SMX have equal rates of cure in the treatment of limited abscess at the TOC visit; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-5.4 to 5.1] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-19.2 to -5.6] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0002, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -12.2, 95% CI 2-sided [-19.1 to -5.4] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

2. Secondary Outcome: Number of Participants Reporting Adverse Events.
Description: Subjects were issued a Memory Aid to record symptoms for 10 days post product administration. At study visits, the staff reviewed the memory aid and elicited as much information as possible about any reported symptoms. Occurrence of adverse events was solicited in the memory aid and during study visits. Reported symptoms, both solicited and unsolicited, were recorded as Adverse Events.
Time Frame: End of Treatment (EOT) (48 hours after completion of therapy); Test of Cure (TOC) (7-10 days after completion of therapy); One Month Follow-up Visit (OMFU)
Population: Participants who received treatment with either clindamycin or TMP/SMX in the cellulitis or larger abscess group and participants who received treatment with either clindamycin, TMP/SMX, or placebo in the limited abscess group.
Measure: Number; unit: participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 259 | 258 | 265 | 261 | 255
participants | 116 | 132 | 119 | 94 | 119

3. Secondary Outcome: Number of Participants Reporting Adverse Events That Are Treatment Limiting.
Description: Participants were issued a Memory Aid to record symptoms for 10 days post product administration. At study visits, the staff reviewed the memory aid and elicited as much information as possible about any reported symptoms. Occurrence of adverse events was solicited in the memory aid and during study visits. Reported symptoms, both solicited and unsolicited, were recorded as Adverse Events. For these results, adverse events that resulted in discontinuation of study treatment for the participant were considered treatment limiting.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 259 | 258 | 265 | 261 | 255
participants | 1 | 0 | 6 | 3 | 4

4. Primary Outcome: Percentage of Participants Achieving Clinical Cure, Defined as Absence of Clinical Failure, in the Intent-to-Treat (ITT) Population.
Description: as for outcome 1
Time Frame: Test of cure (TOC) (7-10 days after completion of therapy)
Population: The ITT population was comprised of all participants enrolled in the trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 264 | 260 | 266 | 263 | 257
percentage of participants | 80.3 [75.2 to 85.4] | 77.7 [72.3 to 83.1] | 83.1 [78.3 to 87.9] | 81.7 [76.8 to 86.7] | 68.9 [62.9 to 74.9]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5200, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-10.2 to 4.9] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7324, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-8.4 to 5.7] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0001, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -14.2, 95% CI 2-sided [-22.0 to -6.4] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0008, Fisher Exact — Adjustments for multiple comparisons were made using a Bonferroni correction; Mean Difference (Final Values) = -12.9, 95% CI 2-sided [-20.8 to -5.0] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

5. Secondary Outcome: Percentage of Participants Achieving Clinical Cure at the End of Treatment (EOT) Visit for the Evaluable Population.
Description: Measures of clinical cure and clinical failure are the same as those defined for the primary efficacy outcome measure.
Time Frame: EOT visit within 48 hours of completion of therapy
Population: The efficacy evaluable population was comprised of all participants who had outcomes determined at the EOT visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 240 | 222 | 231 | 223 | 219
percentage of participants | 89.2 [85.0 to 93.3] | 88.3 [83.8 to 92.7] | 90.9 [87.0 to 94.8] | 94.2 [90.9 to 97.5] | 84.9 [80.0 to 89.9]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; Null hypothesis: Clindamycin and TMP-SMX have equal rates of cure in the treatment of cellulitis/larger abscess; Test type: Superiority or Other; p = 0.7707, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-7.1 to 5.3] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; Null hypothesis: After successful surgical drainage, placebo, Clindamycin, and TMP-SMX have equal rates of cure in the treatment of limited abscess; Test type: Superiority or Other; p = 0.2141, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-2.0 to 8.5] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0593, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-12.4 to 0.5] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0017, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -9.2, 95% CI 2-sided [-15.3 to -3.1] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

6. Secondary Outcome: Percentage of Participants Achieving Clinical Cure at the End of Treatment (EOT) Visit for the Intent-to-Treat (ITT) Population.
Description: Measures of clinical cure and clinical failure are the same as those defined for the primary efficacy outcome measure.
Time Frame: EOT visit within 48 hours of completion of therapy
Population: All participants enrolled in the trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 264 | 260 | 266 | 263 | 257
percentage of participants | 81.1 [76.1 to 86.0] | 75.4 [70.0 to 80.8] | 78.9 [73.9 to 84.0] | 79.8 [74.8 to 84.9] | 72.4 [66.7 to 78.0]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; Null hypothesis: Clindamycin and TMP-SMX have equal rates of cure in the treatment of cellulitis/larger abscess; Test type: Superiority or Other; p = 0.1381, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-13.1 to 1.8] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.8302, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-6.4 to 8.2] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0838, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -6.6, 95% CI 2-sided [-14.3 to 1.1] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0507, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-15.2 to 0.2] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

7. Secondary Outcome: Percentage of Participants Achieving Clinical Cure at the One Month Follow-up (OMFU) Visit for the Evaluable Population.
Description: Measures of clinical cure and clinical failure are the same as those defined for the primary efficacy outcome measure, with one addition. At the OMFU, relapse (the return of the original infection after initial improvement) or recurrence (return of skin infection at original site after cure of original infection) of SSTI was scored as clinical failure.
Time Frame: OMFU visit
Population: The efficacy evaluable population was comprised of all participants who had outcomes determined at the OMFU visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 230 | 225 | 234 | 226 | 218
percentage of participants | 83.9 [78.9 to 88.9] | 78.2 [72.6 to 83.8] | 89.3 [85.1 to 93.5] | 85.0 [80.1 to 89.8] | 73.9 [67.8 to 79.9]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; Null hypothesis: Clindamycin and TMP-SMX have equal rates of cure in the treatment of cellulitis/larger abscess; Test type: Superiority or Other; p = 0.1505, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-13.3 to 1.9] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.1666, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -4.4, 95% CI 2-sided [-10.9 to 2.2] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -15.5, 95% CI 2-sided [-23.0 to -8.0] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0046, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -11.1, 95% CI 2-sided [-19.0 to -3.2] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

8. Secondary Outcome: Percentage of Participants Achieving Clinical Cure at the One Month Follow-up (OMFU) Visit for the Intent-to-Treat (ITT) Population.
Description: as for outcome 7
Time Frame: OMFU visit
Population: All participants enrolled in the trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Number analyzed (Participants) | 264 | 260 | 266 | 263 | 257
percentage of participants | 73.1 [67.6 to 78.6] | 67.7 [61.8 to 73.6] | 78.6 [73.5 to 83.7] | 73.0 [67.4 to 78.6] | 62.6 [56.5 to 68.8]
Statistical Analysis 1: Comparison: Cellulitis or Larger Abscess - Clindamycin vs Cellulitis or Larger Abscess - TMP-SMX; Null hypothesis: Clindamycin and TMP-SMX have equal rates of cure in the treatment of cellulitis/larger abscess; Test type: Superiority or Other; p = 0.1815, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-13.6 to 2.8] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 2: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - TMP-SMX; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.1552, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-13.2 to 2.1] — The mean difference is determined by the cure rate of TMP-SMX minus Clindamycin
Statistical Analysis 3: Comparison: Limited Abscess - Clindamycin vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -15.9, 95% CI 2-sided [-24.0 to -7.8] — The mean difference is determined by the cure rate of Placebo minus Clindamycin
Statistical Analysis 4: Comparison: Limited Abscess - TMP-SMX vs Limited Abscess - Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.0145, Fisher Exact — Adjustments for multiple comparisons were not made for secondary efficacy outcome measures; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-18.7 to -2.0] — The mean difference is determined by the cure rate of Placebo minus TMP-SMX

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected after administration of the first dose of study drug throughout the duration of the follow-up period (35-45 days after enrollment).
Groups:
- Cellulitis or Larger Abscess - Clindamycin: Participants with cellulitis only or abscess > 5 cm in diameter, or with 2 or more sites of skin infection were treated with CLINDA300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children.
- Cellulitis or Larger Abscess - TMP-SMX: Participants with cellulitis only or abscess > 5 cm in diameter, or with 2 or more sites of skin infection were treated with TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children.
- Limited Abscess - Clindamycin: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter were treated with CLINDA300 mg three times daily for adults; 25-30 mg/kg/day divided three times daily for children.
- Limited Abscess - TMP-SMX: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter were treated with TMP-SMX 160/800 mg twice daily for adults; 8-10 mg/kg of TMP, 40-50 mg/kg of SMX twice daily for children.
- Limited Abscess - Placebo: Participants with limited abscess with or without cellulitis less than or equal to 5 cm in diameter were treated with placebo three times daily.
Arm/Group | Cellulitis or Larger Abscess - Clindamycin | Cellulitis or Larger Abscess - TMP-SMX | Limited Abscess - Clindamycin | Limited Abscess - TMP-SMX | Limited Abscess - Placebo
Serious Adverse Events (participants affected / at risk) | 4/264 | 5/260 | 0/266 | 6/263 | 2/257
Other Adverse Events (participants affected / at risk) | 59/264 | 72/260 | 61/266 | 52/263 | 60/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellulitis or Larger Abscess - Clindamycin (N=264) | Cellulitis or Larger Abscess - TMP-SMX (N=260) | Limited Abscess - Clindamycin (N=266) | Limited Abscess - TMP-SMX (N=263) | Limited Abscess - Placebo (N=257)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cellulitis or Larger Abscess - Clindamycin (N=264) | Cellulitis or Larger Abscess - TMP-SMX (N=260) | Limited Abscess - Clindamycin (N=266) | Limited Abscess - TMP-SMX (N=263) | Limited Abscess - Placebo (N=257)
Abscess (Infections and infestations) | 21 (23) | 39 (43) | 13 (13) | 29 (30) | 35 (36)
Cellulitis (Infections and infestations) | 16 (19) | 23 (26) | 3 (3) | 6 (6) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 27 (30) | 28 (29) | 46 (48) | 17 (19) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less